CLINICAL TRIAL: NCT01689857
Title: Phase 4 Study of Scarclinic™ Thin That Treats Surgical Scars.
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of Scarclinic™ Thin in Surgical Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chan-Yeong Heo, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-1004-048-004; 06-2010-049 (Other Grant/Funding Number: ILDONG Pharmaceutical CO. LTD.)
Record Dates: First submitted 2012-09-13; First posted 2012-09-21 (Estimated); Results first posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Hypertrophic Surgical Scar
Keywords: hypertropic scar, Vancouver scar scale, silicon gel sheet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scarclinic™ Thin (Experimental): Scarclinic™ Thin
  Interventions: Device: Scarclinic™ Thin
- Scarclinic™ Normal (Active Comparator): Scarclinic™ Normal
  Interventions: Device: Scarclinic™ Normal

INTERVENTIONS:
Device: Scarclinic™ Thin — Apply Scarclinic™ Thin on the scar and dispense 4 ea.for each participant for 3 month.
  Arms: Scarclinic™ Thin
Device: Scarclinic™ Normal — Apply Scarclinic™ Normal on the scar and dispense 4 ea.for each participant for 3 month.
  Arms: Scarclinic™ Normal

SUMMARY:
Compare the efficacy and safety of Scarclinic™Thin and Scarclinic™ Normal for the treatment of surgical scars.

Participant: 40 Treatment period : 3 months Medical device: Scarclinic™Thin , Scarclinic™ Normal Randomization: Table of random number

DETAILED DESCRIPTION:
For evaluating the efficacy

* The investigator check Vancouver Scar Scale at 1 and 3 month after application to evaluate vascularity, pigmentation, elasticity, height, pain and itchiness
* The participant filled out survey included questions regarding convenience in use at 1 and 3 month after application.

ELIGIBILITY:
Inclusion Criteria:

* Patient who aged more than 18 years and less 55 years
* Patient who has a surgical scar that is not over 3 months after the surgery
* Patient who sign informed consent form for the study

Exclusion Criteria:

* need wound dressing for exudate
* wound infection
* general malaise
* history of mental disorders
* taking anticancer drugs or antiphlogistics or steroid

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ChanYoung Heo, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Bundang-gu, Seongnam-si,Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Seoul National University Bundang hospital. Forty subjects were recruited from May, 2010 to April,2012.
Pre-assignment Details: In this study, we had no run-in period before study was commenced and there were no subjects who drop out before enrollment and randomization to groups.
Groups:
- Scarclinic™ Thin: Scarclinic™ Thin applied on the surgical scar for 12weeks
- Scarclinic™ Normal: Scarclinic™ Normal applied on the surgical scar for 12weeks
Period: Overall Study
Arm/Group | Scarclinic™ Thin | Scarclinic™ Normal
Started | 20 | 20
Completed | 15 | 18
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scarclinic™ Thin | Scarclinic™ Normal | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.90 (10.47) | 36.00 (9.93) | 37.95 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Vancouver Scar Scale Score(VSS) at 3 Months
Description: Scar assessment will be performed at the beginning of the treatment, and at the end of the 3 month when the treatment is completed by using the Vancouver scar scale.VSS assesses 6 variables.
  * vascularity(range from normal(0 point) to purple(3point)
  * pigmentation(range from normal(0 point) to hyper-pigmentation(3point)
  * pliability(range from normal(0 point) to contracture(5point)
  * height (range from flat(0 point) to above 5mm(3point)
  * pain(range from none(0 point) to Require medication(2point)
  * itchiness(range from none(0 point) to Require medication(2point)
  We assess total score that are minimum score is 0 and maximum is 18. The lowest score means the best scar condition.
Time Frame: Baseline and 3 months
Population: All participants for whom Vancouver Scar Scale measurements were recorded at Baseline and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scarclinic™ Thin | Scarclinic™ Normal
Number analyzed (Participants) | 15 | 18
units on a scale | -3.80 (3.02) | -2.61 (2.63)

2. Secondary Outcome: Satisfaction for Serviceability
Description: Satisfaction for serviceability will be performed at the end of the 3 month when the treatment was completed by using Questionaire
Time Frame: the end of the 3 month of the treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Scarclinic™ Thin | Scarclinic™ Normal
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 12/20 | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scarclinic™ Thin (N=20) | Scarclinic™ Normal (N=20)
itching sense (Skin and subcutaneous tissue disorders) | 10 (10) | 8 (8)
redness (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No